CLINICAL TRIAL: NCT01014247
Title: A Randomized, Double-blind, 2-way Crossover, Placebo-controlled Study to Investigate the Influence of a Single-dose of Moxifloxacin on the QTc Interval in Healthy Male and Female Subjects for Positive Control Validation in Selected Centers of the PATENT-1 Trial
Brief Title: Influence of Moxifloxacin on QTc Interval in Healthy Subjects for Positive Control Validation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer HealthCare Pharmaceuticals Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 13796; 2009-012363-34 (EudraCT Number)
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: QTc Evaluation; Electrocardiography
Keywords: Moxifloxacin
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — Single dose of 400 mg
  Arms: Arm 1
Drug: Placebo — Single dose of matching tablet
  Arms: Arm 2

SUMMARY:
The aim of this study is to investigate the effect of moxifloxacin on the QT interval in order to gain information on the validity of results that will be collected during another clinical study testing riociguat in patients with pulmonary arterial hypertension (PATENT-1 study).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18-75 years - Normal ECG Exclusion Criteria:
* Abnormal ECG - Intolerance to fluorochinolones

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
QTc interval at 3 hours | Day 1 of treatment period 1 and 2

SECONDARY OUTCOMES:
Safety variables | Up to last visit of follow up
  Adverse events, clinical laboratory, vital signs, ECG findings
Pharmacokinetic parameters | On different time points
  Cmax, Cmax,norm, tmax

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Melbourne, Victoria, Australia
- Germany (2):
  - Giessen, Hesse
  - Dresden, Saxony
- Singapore, Singapore
- London, United Kingdom